CLINICAL TRIAL: NCT06112496
Title: Effect of Smartphone Addiction on the Myoelectrical Activity of the Sternocleidomastoid Muscle in Adult
Brief Title: Effect of Smartphone Addiction on Myoelectrical Activity of Sternocleidomastoid Muscle in Adult
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Huda Adel Mohammed Hassan, principal investigator, Cairo University
Other Study IDs: P.T.REC/012/004614
Record Dates: First submitted 2023-10-19; First posted 2023-11-01 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Heavy Smart Phone Users

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- smart phone addict
  Interventions: Device: EMG
- smart phone non addict
  Interventions: Device: EMG

INTERVENTIONS:
Device: EMG — Neuro-EMG-Micro, Neurosoft, Ivanovo, Russia, will be used for the assessment of muscle activity for muscles.

SUMMARY:
This study will be conducted to identify the effect of smartphone addiction myoelectrical activity on sternocleidomastoid in adults by measuring The amplitude of EMG signals of the sternocleidomastoid muscle in adults and Root mean square of EMG signals of the sternocleidomastoid muscle in adults

ELIGIBILITY:
Inclusion Criteria:

* Subject's age range from 18-30 years old
* All participants use the same smartphone with a touch screen of 6,7 inches.

Exclusion Criteria:

* Neck pain ( spondylosis, spondylolysis)
* Systemic diseases.
* Spinal deviation

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: smart phone users
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2023-12-16 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Changes in surface electromyographic (EMG) amplitude of sternocleidomastoid muscle | day 1
  change in amplitude measured by EMG device
change in RMS | day 1
  change in root mean square measured by EMG device

CONTACTS AND LOCATIONS:
Locations (1):
- Huda Adel, Cairo, Egypt